CLINICAL TRIAL: NCT00510952
Title: The PERSISTENT Trial: A Prospective Randomized Trial Comparing Insulin Lispro Protamine Suspension to Insulin Glargine in Patients With Type 2 Diabetes on Anti-hyperglycemic Medications
Brief Title: Comparison of Two Basal Insulins for Patients With Type 2 Diabetes on Anti-Hyperglycemic Medications (IOPE)
Acronym: IOPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11813; F3Z-MC-IOPE (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Results first posted 2009-11-03 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — neutral protamine lispro insulin; Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lispro (Experimental): Insulin Lispro protamine suspension: Patient adjusted dose, once daily (QD) or twice daily (BID), injected subcutaneous (SC) x 24 weeks
  Interventions: Drug: Insulin Lispro Protamine Suspension
- Glargine (Active Comparator): Insulin glargine: Patient adjusted dose, once daily (QD), injected subcutaneous (SC) x 24 weeks
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Lispro Protamine Suspension — Patient adjusted dose, once daily (QD) or twice daily (BID), injected subcutaneous (SC) x 24 weeks
  Other Names: Insulin Lispro Protamine Suspension (ILPS); Neutral Protamine Lispro (NPL); Humalog
  Arms: Lispro
Drug: Insulin Glargine — Patient adjusted dose, once daily (QD), injected subcutaneous (SC) x 24 weeks
  Arms: Glargine

SUMMARY:
The purpose of this study is to examine the effectiveness and safety of insulin lispro protamine suspension (ILPS) as compared to insulin glargine as basal insulin therapy in adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus for at least 1 year.
* Are greater than or equal to 18 years old.
* Have been receiving oral antihyperglycemic medications (OAMs), without insulin, for at least 3 months immediately prior to the study and have been on stable doses of at least 2 of the following OAMs for the 6 weeks prior to Visit 1: Metformin- Sulfonylureas-Dipeptidyl peptidase-IV (DPP-IV) inhibitors-Thiazolidinediones (TZDs)
* Have a hemoglobin A1c (HbA1c) greater than or equal to 7.5% and less than or equal to 10.0%, as measured by a central laboratory before Visit 2.
* Body mass index (BMI) greater than or equal to 25 and less than or equal to 45 kg/meter squared.

Exclusion Criteria:

* Have used insulin therapy (outside of pregnancy) any time in the past 2 years, except for short-term treatment of acute conditions, and up to a maximum of 4 weeks.
* Have taken any glucose-lowering medications not included in Inclusion Criterion #3; (for example, acarbose, miglitol, pramlintide, exenatide, repaglinide, or nateglinide) in the past 3 months before Visit 1.
* Have had more than 1 episode of severe hypoglycemia, within 6 months prior to entry into the study, or is currently diagnosed as having hypoglycemia unawareness.
* Have had 2 or more emergency room visits or hospitalizations due to poor glucose control in the past 6 months.
* Are pregnant or intend to become pregnant during the course of the study or are sexually active women of childbearing potential not actively practicing birth control by a method determined by the investigator to be medically acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM-5 PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jonesboro, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntington Park, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Slidell, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
- Brazil (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasília
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fortaleza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Joinville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia, Canada
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce, Puerto Rico

REFERENCES:
- [Result] Strojek K, Shi C, Carey MA, Jacober SJ. Addition of insulin lispro protamine suspension or insulin glargine to oral type 2 diabetes regimens: a randomized trial. Diabetes Obes Metab. 2010 Oct;12(10):916-22. doi: 10.1111/j.1463-1326.2010.01257.x. PMID 20920045
- [Derived] Qu Y, Jacober SJ, Zhang Q, Wolka LL, DeVries JH. Rate of hypoglycemia in insulin-treated patients with type 2 diabetes can be predicted from glycemic variability data. Diabetes Technol Ther. 2012 Nov;14(11):1008-12. doi: 10.1089/dia.2012.0099. PMID 23101951
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lispro | Glargine
Started | 235 | 236
Full Analysis Set (Intent to Treat) | 229 | 229
Completed | 209 | 220
Not Completed | 26 | 16
Not completed — Adverse Event | 1 | 0
Not completed — Entry Criteria Not Met | 3 | 1
Not completed — Lost to Follow-up | 5 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 7 | 4
Not completed — Sponsor Decision | 1 | 0
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Did Not Receive Study Drug | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lispro | Glargine | Total
Number analyzed (Participants) | 229 | 229 | 458
Age Continuous [Mean (Standard Deviation); unit: years] | 58.05 (9.35) | 57.29 (8.99) | 57.67 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 116 | 223
  Male | 122 | 113 | 235
Region of Enrollment [Number; unit: participants]
  Argentina | 13 | 12 | 25
  Brazil | 18 | 19 | 37
  Canada | 20 | 20 | 40
  India | 27 | 31 | 58
  Korea, Republic of | 9 | 13 | 22
  Mexico | 18 | 16 | 34
  Poland | 52 | 50 | 102
  Russian Federation | 30 | 29 | 59
  Spain | 9 | 10 | 19
  United States | 33 | 29 | 62
Race/Ethnicity [Number; unit: participants]
  African | 11 | 14 | 25
  Caucasian | 147 | 142 | 289
  East Asian | 10 | 15 | 25
  Hispanic | 33 | 26 | 59
  Native American | 0 | 1 | 1
  West Asian (Indian sub-continent) | 28 | 31 | 59
Sulfonylurea Group [Number; unit: participants] — Patients with previous sulfonylurea use.
  participants
    Yes | 191 | 190 | 381
    No | 38 | 39 | 77
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 30.69 (5.01) | 31.62 (5.48) | 31.16 (5.27)
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 84.23 (16.83) | 86.05 (18.62) | 85.14 (17.75)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 9.80 (6.45) | 9.90 (6.51) | 9.85 (6.47)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 165.45 (10.04) | 164.62 (10.11) | 165.03 (10.07)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Week Endpoint in Hemoglobin A1c (HbA1c)
Time Frame: Baseline, 24 Weeks
Population: Number of randomized patients who received at least one dose of study drug and had at least one post-baseline measurement. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: percent of HbA1c
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 225 | 226
percent of HbA1c
  Baseline | 8.70 (0.06) | 8.69 (0.06)
  Change from Baseline | -1.46 (0.07) | -1.41 (0.07)
Statistical Analysis 1: Comparison: Lispro vs Glargine; Hypothesis: Basal analog insulin lispro protamine suspension, injected once or twice daily is noninferior to basal analog insulin glargine, injected once a day, with regard to glycemic control as measured by change in HbA1c from baseline to 24 week endpoint (last observation carried forward); Test type: Non-Inferiority or Equivalence — Noninferiority margin was 0.4%; p = 0.551, ANCOVA — P-value for Change from Baseline; ANCOVA Model: Variable = Treatment + Baseline + Country + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.05, 95% CI [-0.21 to 0.11] — The two-sided 95% confidence interval is for the Least Squares Mean difference between the two treatments (Insulin Lispro Protamine Suspension minus Glargine)

2. Secondary Outcome: Actual and Change From Baseline to 12 Week and 24 Week Endpoint in HbAlc Value
Time Frame: Baseline, 12 Weeks, 24 Weeks
Population: Number of randomized patients who received at least one dose of study drug and had at least one post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percent hemoglobin
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 229 | 229
percent hemoglobin
  Baseline (n= 225, n= 226) | 8.70 (0.06) | 8.69 (0.06)
  Week 12 HbA1c (n=213, n=220) | 7.30 (0.07) | 7.36 (0.07)
  Week 12 Change from Baseline (n=213, n=220) | -1.36 (0.07) | -1.30 (0.07)
  Week 24 HbA1c (n=206, n=218) | 7.15 (0.07) | 7.24 (0.07)
  Week 24 Change from Baseline (n=206, n=218) | -1.52 (0.07) | -1.43 (0.07)
Statistical Analysis 1: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.427, ANCOVA — P-value for Week 12 HbA1c; ANCOVA Model: Variable = Treatment + Baseline + Country + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.06, 95% CI [-0.21 to 0.09] — The two-sides 95% confidence interval is for the Least Squares Mean difference between the two treatments (Insulin Lispro Protamine Suspension minus Glargine)
Statistical Analysis 2: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.427, ANCOVA — P-value for Week 12 Change from Baseline; ANCOVA Model: Variable = Treatment + Baseline + Country + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.06, 95% CI [-0.21 to 0.09] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.254, ANCOVA — P-value for Week 24 HbA1c; ANCOVA Model: Variable = Treatment + Baseline + Country + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.09, 95% CI [-0.25 to 0.07] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.254, ANCOVA — P-value for Week 24 Change from Baseline; ANCOVA Model: Variable = Treatment + Baseline + Country + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.09, 95% CI [-0.25 to 0.07] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Patients With HbAlc Less Than 7.0 Percent and HbAlc Less Than or Equal to 6.5 Percent at Endpoint
Description: Percentage of patients achieving Hemaglobin A1c (HbA1c) targets of less than 7% and less than or equal to 6.5% at endpoint.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 226 | 226
percentage of participants
  HbA1c <7.0% | 43.8 | 41.2
  HbA1c ≤6.5% | 24.8 | 21.7
Statistical Analysis 1: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.634, Fisher Exact — P-value for HbA1c <7.0%
Statistical Analysis 2: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.504, Fisher Exact — P-value for HbA1c ≤6.5%

4. Secondary Outcome: Glycemic Variability at Endpoint
Description: Glycemic variability was measured by standard deviation (SD) value of fasting blood glucose as measured by intra-patient glycemic variability (determined by the 7-point self-monitoring blood glucose (SMBG) profiles at endpoint) based on the actual morning pre-meal blood glucose.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 228 | 229
millimoles per liter (mmol/L) | 1.01 (0.72) | 0.94 (0.71)
Statistical Analysis 1: Comparison: Lispro vs Glargine; Hypothesis: Insulin lispro protamine suspension is noninferior to glargine at actual morning pre-meal at endpoint; Test type: Non-Inferiority or Equivalence — Noninferiority margin of 0.8 millimoles per liter (mmol/L); p = 0.323, ANOVA; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group; Mean Difference (Net) = 0.06, 95% CI [-0.06 to 0.19] — The two-sided 95% confidence interval is for the Least Squares Mean difference between the two treatment groups (Insulin Lispro Protamine Suspension minus Glargine)

5. Secondary Outcome: 7-Point Self-Monitored Blood Glucose (SMBG) Profile at Endpoint
Description: Actual measurements and daily mean blood glucose levels at endpoint.
Time Frame: 24 weeks
Population: Number of randomized patients who received at least one dose of study drug and at least one post-baseline measurement. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 226 | 226
millimoles per liter (mmol/L)
  Actual Morning Pre-Meal | 6.47 (1.40) | 6.33 (1.36)
  Actual Morning Postprandial Meal | 8.64 (2.48) | 9.00 (2.55)
  Actual Midday Pre-Meal | 6.93 (2.11) | 7.16 (2.07)
  Actual Midday Postprandial Meal | 9.09 (2.52) | 9.17 (2.50)
  Actual Evening Pre-Meal | 7.50 (2.06) | 7.54 (2.02)
  Actual Evening Postprandial Meal | 9.19 (2.84) | 9.29 (2.54)
  Actual 0300 Hours | 6.79 (2.05) | 7.00 (2.21)
  Daily Mean 7-Point SMBG | 7.79 (1.82) | 7.96 (1.74)
  Daily Mean Pre-Meal | 6.99 (1.77) | 7.04 (1.55)
  Daily Mean Postprandial Meal | 8.96 (2.25) | 9.18 (2.20)
  Daily Mean Morning+Evening Pre-Meal | 6.99 (1.51) | 6.93 (1.41)
Statistical Analysis 1: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.302, ANOVA — P-value for Actual Morning Pre-Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 2: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.144, ANOVA — P-value for Actual Morning Postprandial Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 3: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.279, ANOVA — P-value for Actual Midday Pre-Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 4: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.928, ANOVA — P-value for Actual Midday Postprandial Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 5: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.918, ANOVA — P-value for Actual Evening Pre-Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 6: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.875, ANOVA — P-value for Actual Evening Postprandial Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 7: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.316, ANOVA — P-value for Actual 0300 Hours; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 8: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.389, ANOVA — P-value for Daily Mean 7-Point SMBG; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 9: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.836, ANOVA — P-value for Daily Mean Pre-Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 10: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.394, ANOVA — P-value for Daily Mean Postprandial Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group
Statistical Analysis 11: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.609, ANOVA — P-value for Daily Mean Morning+Evening Pre-Meal; ANOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group

6. Secondary Outcome: Number of Participants With Self-Reported Hypoglycemic Episodes (Including All, Nocturnal, and Severe Hypoglycemia) Overall
Description: Overall: any time after randomization. Hypoglycemic: any time patient experienced sign/symptom associated with hypoglycemia, or had old Roche blood glucose level <7 mg/dL. Nocturnal: any hypoglycemic event that occurred between bedtime and waking. Severe Hypoglycemia: event with symptoms consistent with neuroglycopenia in which patient requires assistance, and is associated with either a Roche blood glucose value <2.8 millimoles/liter or prompt recovery after oral carbohydrate, glucagon, or intravenous glucose.
Time Frame: Baseline to 24 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 229 | 229
participants
  All Hypoglycemic Episodes | 168 | 160
  Nocturnal Hypoglycemic Episodes | 114 | 87
  Severe Hypoglycemic Episodes | 9 | 2
Statistical Analysis 1: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.468, Fisher Exact — P-value for All Hypoglycemic Episodes
Statistical Analysis 2: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.011, Fisher Exact — P-value for Nocturnal Hypoglycemic Episodes
Statistical Analysis 3: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.036, Fisher Exact — P-value for Severe Hypoglycemic Episodes

7. Secondary Outcome: 1-Year Adjusted Rates of Self-Reported Hypoglycemic Episodes (Including All, Nocturnal, and Severe) Overall
Description: Overall: any time after randomization. Hypoglycemic: any time patient experienced sign/symptom associated with hypoglycemia, or had old Roche blood glucose level <7 mg/dL. Nocturnal: any hypoglycemic event that occurred between bedtime and waking. Severe: event with symptoms consistent with neuroglycopenia in which patient requires assistance, and is associated with: a Roche blood glucose value <2.8 mmol/L or prompt recovery after oral carbohydrate, glucagon, or IV glucose. 1-year adjusted rate=(total number of episodes between 2 time intervals/number of days between intervals) X 365.25 days.
Time Frame: Baseline to 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hypoglycemic event per 1 year
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 229 | 229
hypoglycemic event per 1 year
  Hypoglycemic Rate | 24.16 (28.78) | 22.95 (30.87)
  Nocturnal Hypoglycemic Rate | 6.08 (10.62) | 4.08 (9.40)
  Severe Hypoglycemic Rate | 0.11 (0.58) | 0.02 (0.21)
Statistical Analysis 1: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.316, ANOVA — P-value for Hypoglycemic Rate; Nonparametric ANOVA Model: Rank of Variable=Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group. Hypoglycemic Rate (1 year) was used
Statistical Analysis 2: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p < 0.001, ANOVA — P-Value for Nocturnal Hypoglycemic Rate; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.102, ANOVA — P-value for Severe Hypoglycemic Rate; [statistical method as in outcome 7, analysis 1]

8. Secondary Outcome: 30-Day Adjusted Rates of Self-Reported Hypoglycemic Episodes (Including All, Nocturnal, and Severe) Overall
Description: Overall: any time after randomization. Hypoglycemic: any time patient experienced sign/symptom associated with hypoglycemia, or had old Roche blood glucose level <7 mg/dL. Nocturnal: any hypoglycemic event that occurred between bedtime and waking. Severe: event with symptoms consistent with neuroglycopenia in which patient requires assistance, and is associated with: a Roche blood glucose value <2.8 mmol/L or prompt recovery after oral carbohydrate, glucagon, or IV glucose. 30-day adjusted rate=(total number of episodes between 2 time intervals/number of days between intervals) X 30 days.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hypoglycemic events per 30 days
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 229 | 229
hypoglycemic events per 30 days
  Hypoglycemic Rate | 1.98 (2.36) | 1.88 (2.54)
  Nocturnal Hypoglycemic Rate | 0.50 (0.87) | 0.34 (0.77)
  Severe Hypoglycemic Rate | 0.01 (0.05) | 0.00 (0.02)

9. Secondary Outcome: Change in Absolute Body Weight (kg) From Baseline to 24 Week Endpoint
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 229 | 229
kilograms (kg)
  Baseline | 84.23 (16.83) | 86.05 (18.62)
  Change from Baseline | 1.04 (3.45) | 1.07 (3.25)
Statistical Analysis 1: Comparison: Lispro vs Glargine; Hypothesis: insulin lispro protamine suspension is noninferior to glargine with regard to change in absolute body weight from baseline to endpoint; Test type: Non-Inferiority or Equivalence — Noninferiority margin of 1.5 kilograms (kg); p = 0.975, ANCOVA — P-value for Change from Baseline; ANCOVA Model: Variable = Treatment + Baseline + Country + Baseline HbA1c + Baseline Sulfonylurea Group; Mean Difference (Net) = -0.01, 95% CI [-0.61 to 0.59] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Total Daily Insulin Dose (Units) at Endpoint
Description: Insulin dose at endpoint was analyzed by 24-hour total daily insulin (units).
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units of insulin
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 229 | 228
Units of insulin | 33.28 (21.84) | 30.85 (20.46)
Statistical Analysis 1: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.031, ANCOVA; ANCOVA Model: Variable = Treatment + Country + Baseline HbA1c + Baseline Sulfonylurea Group + Change in HbA1c from Baseline

11. Secondary Outcome: Total Daily Insulin Dose Per Body Weight (Units/Kilograms) at Endpoint
Description: Insulin dose at endpoint was analyzed by 24-hour total daily insulin per body weight (units/kilograms).
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units of insulin/kilograms (U/kg)
Arm/Group | Lispro | Glargine
Number analyzed (Participants) | 229 | 228
Units of insulin/kilograms (U/kg) | 0.39 (0.24) | 0.35 (0.20)
Statistical Analysis 1: Comparison: Lispro vs Glargine; Test type: Superiority or Other; p = 0.015, ANCOVA; [statistical method as in outcome 10, analysis 1]

ADVERSE EVENTS:
Arm/Group | Lispro | Glargine
Serious Adverse Events (participants affected / at risk) | 4/229 | 10/229
Other Adverse Events (participants affected / at risk) | 100/229 | 109/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lispro (N=229) | Glargine (N=229)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Retinal ischaemia (Eye disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lispro (N=229) | Glargine (N=229)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 8 (8)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Chest pain (General disorders) | 3 (3) | 4 (6)
Fatigue (General disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 4 (5) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4)
Influenza (Infections and infestations) | 8 (10) | 11 (12)
Nasopharyngitis (Infections and infestations) | 10 (10) | 17 (17)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 8 (10) | 5 (5)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (7)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 6 (6)
Headache (Nervous system disorders) | 15 (25) | 12 (22)
Paraesthesia (Nervous system disorders) | 4 (5) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (5) | 5 (5)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 6 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 6 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days